CLINICAL TRIAL: NCT02387138
Title: A Phase I Trial Assessing Several Schedules of Oral S-1 in Combination With a Fixed Dose of Oxaliplatin and Irinotecan in Patients With Advanced or Metastatic Digestive Adenocarcinoma as First- or Second-line Treatment
Brief Title: A Trial Assessing Several Schedules of Oral S-1 in Combination With a Fixed Dose of Oxaliplatin and Irinotecan
Acronym: SIRINOX
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Institut du Cancer de Montpellier - Val d'Aurelle (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ICM2013/47
Record Dates: First submitted 2015-03-03; First posted 2015-03-12 (Estimated); Last update posted 2019-08-22 (Actual); Status verified 2017-08

CONDITIONS: Digestive Cancer
MeSH Terms: conditions — Gastrointestinal Neoplasms | interventions — S 1 (combination); Irinotecan; Oxaliplatin; Granulocyte Colony-Stimulating Factor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- SIRINOX (Experimental): S-1: Administered orally twice daily from day 1 for 7 consecutive days followed by a 7-day recovery period in a 14-day cycle.
  The starting dose of S-1 will be two levels below the recommended dose defined in SIRI (20 mg/m² BID minimum) with a cohort dose escalation by 5 mg/m² increments (5 dose levels).
  Irinotecan : fixed dose of 180 mg/m² IV over 90 minutes on d1 of every cycle Oxaliplatin : fixed dose of 85 mg/m² over 120 minutes on d1 of every cycle G-csf : d8 to d13 systematically
  Interventions: Drug: S-1; Drug: Irinotecan; Drug: Oxaliplatin; Other: G-csf

INTERVENTIONS:
Drug: S-1 — S-1: Administered orally twice daily from day 1 for 7 consecutive days followed by a 7-day recovery period in a 14-day cycle.
  The starting dose of S-1 will be two levels below the recommended dose defined in SIRI (20 mg/m² BID minimum) with a cohort dose escalation by 5 mg/m² increments (5 dose levels).
Drug: Irinotecan — Irinotecan : fixed dose of 180 mg/m² IV over 90 minutes on d1 of every cycle
Drug: Oxaliplatin — Oxaliplatin : fixed dose of 85 mg/m² over 120 minutes on d1 of every cycle
Other: G-csf — G-csf : d8 to d13 systematically

SUMMARY:
This study is to determine the Maximal Tolerated Dose (MTD), the Dose Limitant Toxicities (DLTs) and the safety profile of S-1 combined with fixed doses of Irinotecan (SIRI schedule) and fixed doses of Irinotecan and Oxaliplatin (SIRINOX schedule).

DETAILED DESCRIPTION:
Given the therapeutic potential and reduced toxicity advantages of S-1 compared with other fluoropyrimidines, this trial assessing S-1 with Oxaliplatin plus Irinotecan is warranted for future investigations (Phase II-III). The primary objectives are to determine the Maximal Tolerated Dose (MTD), the Dose Limitant Toxicities (DLTs) and the safety profile of S-1 combined with fixed doses of Irinotecan (SIRI schedule) and fixed doses of Irinotecan and Oxaliplatin (SIRINOX schedule).

ELIGIBILITY:
Inclusion Criteria:

* Male or female ≥ 18 years old
* Histologically confirmed diagnosis of advanced or metastatic digestive adenocarcinoma (gastroesophageal adenocarcinoma, colorectal adenocarcinoma, pancreatic adenocarcinoma, cholangiocarcinoma, hepatocarcinoma)
* Metastatic or advanced disease not eligible for curative surgery
* No active biliary obstruction
* Previous adjuvant chemotherapy is allowed. It must be completed at least 6 months before the start of the study treatment
* First line chemotherapy is allowed (excluding chemotherapy with Capecitabine or 5 FU or Irinotecan or Oxaliplatin). Previous Oxaliplatin is allowed in patients receiving SIRI
* A four-week washout period since prior treatment
* One or more measurable metastatic lesions
* ECOG status ≤ 1
* Total bilirubin ≤ 1.5 Upper limit of normal (ULN), ALT or AST ≤ 2.5 ULN (or < 5 in case of liver impairment)
* Haemoglobin ≥ 10 g/dL, neutrophils ≥ 1,500/mm3, platelets ≥ 100,000/mm3 and white blood cells > 3000 /mm3
* Lipase < 1.5 ULN, serum creatinine ≤ 1.5 ULN
* Negative pregnancy test in women of childbearing potential
* Use of an effective contraceptive method during the whole treatment and up to 3 months after the completion of treatment
* Life expectancy > 3 months
* Informed consent form (ICF) signed prior to any study specific procedures
* Patients must be affiliated to a Social Security System

Exclusion Criteria:

* History of previous treatment with Oxaliplatin except for SIRI, Irinotecan, 5 FU or Capecitabine as first-line chemotherapy
* Peripheral sensory neuropathy ≥ grade 2 at the time of signing the ICF
* Known central nervous system metastases
* Unique bone metastasis
* History or presence of other cancer within the past 5 years (except curatively treated non-melanoma skin cancer)
* Patients with a known deficiency of the enzyme dihydropyrimidine dehydrogenase (DPD), as well as patients who, within the previous four weeks, have been treated with a medicine that inhibits this enzyme
* Patients with rare hereditary problems of galactose intolerance, lactase deficiency or glucose or galactose malabsorption
* Malabsorption syndrome or disease significantly affecting gastro-intestinal function
* Patient with dysphagia or inability to swallow the tablets
* Inflammatory bowel disease with chronic diarrhoea (Grade ≥ 2 NCI CTC V4.03)
* History of organ transplantation with use of immunosuppression therapy
* Concomitant severe infection (> grade 2 NCI.CTCAE v4.03) or major organ failure
* Active cardiac disease, angina pectoris or myocardial infarction in the last 6 months
* Renal disease
* Unstable diabetes
* Creatinine clearance < 50 ml/min calculated using the MDRD formula
* Pregnant or breastfeeding women
* Participation in another clinical trial within 30 days prior to study entry
* Psychological, social, geographical or any other condition that would preclude study compliance (treatment administration and study follow-up)
* Legal incapacity or physical, psychological or mental status interfering with the patient's ability to sign the informed consent or to terminate the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2014-04 (Actual); Primary Completion 2018-06 (Actual); Study Completion 2018-09 (Actual)

PRIMARY OUTCOMES:
Dose limiting toxicities | up to 5 years
  Dose limiting toxicities occurring during the first two administered cycles.

CONTACTS AND LOCATIONS:
Overall Officials: SAMALIN Emmanuelle, MD, Principal Investigator — Institut regional du Cancer Montpellier
Locations (1):
- Institut du Cancer de Montpellier - Val d'Aurelle, Montpellier, France